CLINICAL TRIAL: NCT01185080
Title: A Double-blind, Placebo Controlled, Randomised, Parallel Group Phase IIa Study to Investigate the Efficacy, Tolerability, and Safety of Different Dosing Regimens of AZD8848 Administered Intranasally to Seasonal Allergic Rhinitis Patients Out of Pollen Season in a Nasal Allergen Challenge Model
Brief Title: Efficacy Study in Allergic Rhinitis Patients After Intranasal Administration of AZD8848
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0540C00014; 2010-020747-13 (EudraCT Number)
Record Dates: First submitted 2010-08-11; First posted 2010-08-19 (Estimated); Results first posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2015-12

CONDITIONS: Allergic Rhinitis
Keywords: AZD8848; allergic rhinitis; efficacy; tolerability; safety; nasal symptoms
MeSH Terms: conditions — Rhinitis, Allergic | interventions — AZD8848

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1. AZD8848 (Experimental): 20 μg AZD8848 three times weekly
  Interventions: Drug: AZD8848
- 2. Placebo (Placebo Comparator): Placebo three times weekly
  Interventions: Drug: Placebo
- 3. AZD8848 and placebo (Experimental): 60 μg AZD8848 once weekly and placebo twice weekly
  Interventions: Drug: AZD8848 and placebo

INTERVENTIONS:
Drug: AZD8848 — Nasal spray solution, intranasal, three times weekly for one month
  Arms: 1. AZD8848
Drug: Placebo — Nasal spray solution, intranasal, three times weekly for one month
  Arms: 2. Placebo
Drug: AZD8848 and placebo — Nasal spray solution, intranasal, three times weekly for one month
  Arms: 3. AZD8848 and placebo

SUMMARY:
The primary purpose of this study is to investigate effect, tolerability and safety of different dosing regimens of AZD8848 administered intranasally to seasonal allergic rhinitis patients out of season in an allergen challenge model.

DETAILED DESCRIPTION:
A double-blind, placebo controlled, randomised, parallel group phase IIa study to investigate the efficacy, tolerability, and safety of different dosing regimens of AZD8848 administered intranasally to seasonal allergic rhinitis patients out of pollen season in a nasal allergen challenge model

ELIGIBILITY:
Inclusion Criteria:

* Seasonal allergic rhinitis patients out of pollen season
* Have a history and presence of birch and/or timothy grass pollen induced seasonal allergic rhinitis for at least the previous 2 years (verified by a positive skin prick test)
* Patients with need of treatment for their nasal symptoms during the pollen season

Exclusion Criteria:

* Symptomatic perennial allergic or non-allergic rhinitis
* Family history of autoimmune disease A history of asthma

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lennart Greiff, MD, PhD, Principal Investigator — Lund University Hospital, Sweden; Sam Lindgren, MD, PhD, Study Director — AstraZeneca R&D Lund, Sweden
Locations (2):
- Sweden (2):
  - Research Site, Lund, Malmohus Lan
  - Research Site, Helsingborg

REFERENCES:
- [Derived] Greiff L, Ahlstrom-Emanuelsson C, Alenas M, Almqvist G, Andersson M, Cervin A, Dolata J, Lindgren S, Martensson A, Young B, Widegren H. Biological effects and clinical efficacy of a topical Toll-like receptor 7 agonist in seasonal allergic rhinitis: a parallel group controlled phase IIa study. Inflamm Res. 2015 Nov;64(11):903-15. doi: 10.1007/s00011-015-0873-2. Epub 2015 Sep 5. PMID 26342289
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=192&filename=D0540C00014_Study_Synopsis.pdf
- See also: Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=192&filename=AZD8848StudyD0540C00014ARCTIC-CSP_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 93 patients enrolled in the study, who 83 of them were randomized. Of the 10 patients who were not randomized, 3 patients due to "patient decision" and 7 patients due to "Eligibility criteria not fulfilled" were not randomized.
Groups:
- AZD8848 20 μg x3: 20 μg AZD8848 three times weekly
- Placebo: Placebo three times weekly
- AZD8848 60 μg: 60 μg AZD8848 once weekly and placebo twice weekly
Period: Overall Study
Arm/Group | AZD8848 20 μg x3 | Placebo | AZD8848 60 μg
Started | 50 | 16 | 17
Completed | 49 | 15 | 16
Not Completed | 1 | 1 | 1
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Personal reasons | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD8848 20 μg x3 | Placebo | AZD8848 60 μg | Total
Number analyzed (Participants) | 50 | 16 | 17 | 83
Age, Continuous [Mean (Full Range); unit: years] | 29.7 [18 to 53] | 28.8 [20 to 46] | 31.0 [19 to 47] | 29.8 [18 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 2 | 10
  Male | 44 | 14 | 15 | 73

OUTCOME MEASURES:

1. Primary Outcome: Mean of Reflective (10 Min) Total Nasal Symptom Score (TNSS)
Description: Mean of Reflective Total Nasal Symptom Score (absolute values) for symptoms over the last 10 minutes after allergen challenge, collected during clinic visits. The Mean is calculated over the Allergen challenge period, which is a seven day period. Each individual symptom is scored 0 to 3, which 0 = Absence of symptoms, 1 = Mild symptoms, 2 = Moderate symptoms and 3 = Severe symptoms. The scores of each individual symptom (runny nose, blocked nose and the maximum score of nasal itching or sneezing) will be added together to give a TNSS of 0 to 9. TNSS Score 0 indicates better outcome and TNSS score 9 indicates worse outcome.
  Allergen challenge period starts 24 hrs post last dose (visit 15). Number of Participants Analyzed is based on all patients with evaluable efficacy and/or biomarker data from the challenge period (Visit 15).
Time Frame: During 1st day to 7th day of Allergen challenge period.
Measure: Least Squares Mean (Full Range); unit: Scores on a scale
Arm/Group | AZD8848 20 μg x3 | Placebo | AZD8848 60 μg
Number analyzed (Participants) | 50 | 15 | 16
Scores on a scale | 4.52 [1.43 to 7.71] | 4.97 [2.86 to 6.43] | 4.69 [3.14 to 7.00]

2. Primary Outcome: Mean of Reflective (10 Min) Total Nasal Symptom Score (TNSS)
Description: Mean of Reflective Total Nasal Symptom Score (absolute values) for symptoms over the last 10 minutes after allergen challenge, collected during clinic visits. The Mean is calculated over 4th day to 7th day of the Allergen challenge period. Each individual symptom is scored 0 to 3, which 0 = Absence of symptoms, 1 = Mild symptoms, 2 = Moderate symptoms and 3 = Severe symptoms. The scores of each individual symptom (runny nose, blocked nose and the maximum score of nasal itching or sneezing) will be added together to give a TNSS of 0 to 9. TNSS Score 0 indicates better outcome and TNSS score 9 indicates worse outcome. Allergen challenge period starts 24 hrs post last dose.
  Number of Participants Analyzed is based on all patients with evaluable efficacy and/or biomarker data from the challenge period (Visit 15).
Time Frame: During 4th day to 7th day of Allergen challenge period.
Measure: Least Squares Mean (Full Range); unit: Scores on a scale
Arm/Group | AZD8848 20 μg x3 | Placebo | AZD8848 60 μg
Number analyzed (Participants) | 49 | 15 | 16
Scores on a scale | 4.45 [1.25 to 8.25] | 5.36 [3.25 to 8.00] | 4.42 [2.75 to 7.50]

3. Primary Outcome: Mean of Morning Measurements of Reflective (12 Hrs) Total Nasal Symptom Score (TNSS)
Description: Mean of morning measurements of Reflective Total Nasal Symptom Score (absolute values) of symptoms over the last 12 hours during allergen challenge, collected in patient diary. The Mean is calculated over the evening of the 1st day to the morning of 8th day of the Allergen challenge period. Each individual symptom is scored 0 to 3, which 0 = Absence of symptoms, 1 = Mild symptoms, 2 = Moderate symptoms and 3 = Severe symptoms. The scores of each individual symptom (runny nose, blocked nose and the maximum score of nasal itching or sneezing) will be added together to give a TNSS of 0 to 9. TNSS Score 0 indicates better outcome and TNSS score 9 indicates worse outcome.
  Allergen challenge period starts 24 hrs post last dose. Number of Participants Analyzed is based on all patients with evaluable efficacy and/or biomarker data from the challenge period (Visit 15).
Time Frame: During evening of the 1st day to the morning of the 8th day of Allergen challenge period.
Measure: Least Squares Mean (Full Range); unit: Scores on a scale
Arm/Group | AZD8848 20 μg x3 | Placebo | AZD8848 60 μg
Number analyzed (Participants) | 50 | 14 | 16
Scores on a scale | 1.81 [0.286 to 4.14] | 2.14 [0.286 to 3.57] | 1.48 [0.143 to 3.29]

4. Primary Outcome: Mean of Evening Measurements of Reflective (12 Hrs) Total Nasal Symptom Score (TNSS)
Description: Mean of evening measurements of Reflective Total Nasal Symptom Score (absolute values) of symptoms over the last 12 hours during allergen challenge, collected in patient diary. The Mean is calculated over the evening of the 1st day to the morning of 8th day of the Allergen challenge period. Each individual symptom is scored 0 to 3, which 0 = Absence of symptoms, 1 = Mild symptoms, 2 = Moderate symptoms and 3 = Severe symptoms. The scores of each individual symptom (runny nose, blocked nose and the maximum score of nasal itching or sneezing) will be added together to give a TNSS of 0 to 9. TNSS Score 0 indicates better outcome and TNSS score 9 indicates worse outcome.
  Allergen challenge period starts 24 hrs post last dose. Number of Participants Analyzed is based on all patients with evaluable efficacy and/or biomarker data from the challenge period (Visit 15).
Time Frame: During the evening of the 1st day to the morning of the 8th day of Allergen challenge period.
Measure: Least Squares Mean (Full Range); unit: Scores on a scale
Arm/Group | AZD8848 20 μg x3 | Placebo | AZD8848 60 μg
Number analyzed (Participants) | 50 | 14 | 16
Scores on a scale | 2.06 [0.143 to 4.71] | 2.32 [0 to 4.57] | 1.96 [0.143 to 4.43]

5. Primary Outcome: Mean of Peak Nasal Inspiratory Flow (PNIF) (10 Min)
Description: Mean of Peak Nasal Inspiratory Flow (absolute values) recorded immediately after TNSS scoring (recall period 10 min), during Allergen challenge period. The Mean is calculated over the Allergen challenge period, which is a seven day period. The patient will breathe out as much as he can. Then a mask (Portable Inspiratory Flow Meter) will be placed over the nose and mouth and the patient will inspire forcefully through the nose while the lips remain tightly closed. The highest PNIF (L/minute) out of 3 measurements will be recorded.
  Allergen challenge period starts 24 hrs post last dose. Number of Participants Analyzed is based on all patients with evaluable efficacy and/or biomarker data from the challenge period (Visit 15).
Time Frame: During 1st day to 7th day of Allergen challenge period.
Measure: Least Squares Mean (Full Range); unit: L/min
Arm/Group | AZD8848 20 μg x3 | Placebo | AZD8848 60 μg
Number analyzed (Participants) | 50 | 15 | 16
L/min | 117 [37.9 to 197] | 127 [67.0 to 214] | 129 [50.0 to 243]

6. Primary Outcome: Mean of Peak Nasal Inspiratory Flow (PNIF) (10 Min)
Description: Mean of Peak Nasal Inspiratory Flow (absolute values) recorded immediately after TNSS scoring (recall period 10 min), during Allergen challenge period. The Mean is calculated over 4th day to 7th day of the Allergen challenge period. The patient will breathe out as much as he can. Then a mask (Portable Inspiratory Flow Meter) will be placed over the nose and mouth and the patient will inspire forcefully through the nose while the lips remain tightly closed. The highest PNIF (L/minute) out of 3 measurements will be recorded.
  Allergen challenge period starts 24 hrs post last dose. Number of Participants Analyzed is based on all patients with evaluable efficacy and/or biomarker data from the challenge period (Visit 15).
Time Frame: During 4th day to 7th day of Allergen challenge period.
Measure: Least Squares Mean (Full Range); unit: L/min
Arm/Group | AZD8848 20 μg x3 | Placebo | AZD8848 60 μg
Number analyzed (Participants) | 49 | 15 | 16
L/min | 121 [37.5 to 200] | 128 [77.5 to 220] | 135 [52.5 to 245]

7. Primary Outcome: Mean of Morning Measurements of Peak Nasal Inspiratory Flow (PNIF) (12 Hrs)
Description: Mean of morning measurements of Peak Nasal Inspiratory Flow (absolute values) of symptoms over the last 12 hours during allergen challenge, collected in patient diary. The Mean is calculated over the evening of the 1st day to the morning of 8th day of the Allergen challenge period. The patient will breathe out as much as he can. Then a mask (Portable Inspiratory Flow Meter) will be placed over the nose and mouth and the patient will inspire forcefully through the nose while the lips remain tightly closed. The highest PNIF (L/minute) out of 3 measurements will be recorded.
  Allergen challenge period starts 24 hrs post last dose. Number of Participants Analyzed is based on all patients with evaluable efficacy and/or biomarker data from the challenge period (Visit 15).
Time Frame: During evening of the 1st day to the morning of the 8th day of Allergen challenge period.
Measure: Least Squares Mean (Full Range); unit: L/min
Arm/Group | AZD8848 20 μg x3 | Placebo | AZD8848 60 μg
Number analyzed (Participants) | 50 | 14 | 16
L/min | 136 [51.4 to 237] | 148 [84.3 to 237] | 148 [71.4 to 234]

8. Primary Outcome: of Evening Measurements of Peak Nasal Inspiratory Flow (PNIF) (12 Hrs)
Description: Mean of evening measurements of Peak Nasal Inspiratory Flow (absolute values) of symptoms over the last 12 hours during allergen challenge, collected in patient diary. The Mean is calculated over the evening of the 1st day to the morning of 8th day of the Allergen challenge period. The patient will breathe out as much as he can. Then a mask (Portable Inspiratory Flow Meter) will be placed over the nose and mouth and the patient will inspire forcefully through the nose while the lips remain tightly closed. The highest PNIF (L/minute) out of 3 measurements will be recorded.
  Allergen challenge period starts 24 hrs post last dose. Number of Participants Analyzed is based on all patients with evaluable efficacy and/or biomarker data from the challenge period (Visit 15).
Time Frame: During evening of the 1st day to the morning of the 8th day of Allergen challenge period.
Measure: Least Squares Mean (Full Range); unit: L/min
Arm/Group | AZD8848 20 μg x3 | Placebo | AZD8848 60 μg
Number analyzed (Participants) | 50 | 14 | 16
L/min | 145 [52.9 to 222] | 149 [71.4 to 253] | 147 [68.6 to 251]

9. Secondary Outcome: Absolute Mean Value of Instantaneous Total Nasal Symptom Score (TNSS)
Description: Absolute mean value of Instantaneous Total Nasal Symptom Score (TNSS) for pre-dose symptoms on visit 2, during treatment period. Treatment period is one month, which starts at visit 2 and ends at visit 14. Each individual symptom is scored 0 to 3, which 0 = Absence of symptoms, 1 = Mild symptoms, 2 = Moderate symptoms and 3 = Severe symptoms. The scores of each individual symptom (runny nose, blocked nose and the maximum score of nasal itching or sneezing) will be added together to give a TNSS of 0 to 9. TNSS Score 0 indicates better outcome and TNSS score 9 indicate worse outcome.
  Number of Participants Analyzed is based on all patients with evaluable efficacy and/or biomarker data at visit 2.
Time Frame: Pre-dose on visit 2 (baseline)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | AZD8848 20 μg x3 | Placebo | AZD8848 60 μg
Number analyzed (Participants) | 50 | 16 | 17
Scores on a scale | 0.38 (0.697) | 0.75 (1.291) | 0.35 (0.493)

10. Secondary Outcome: Absolute Mean Value of Instantaneous Total Nasal Symptom Score (TNSS)
Description: Absolute mean value of Instantaneous Total Nasal Symptom Score (TNSS) for pre-dose symptoms on visit11, during treatment period. Treatment period is one month, which starts at visit 2 and ends at visit 14. Each individual symptom is scored 0 to 3, which 0 = Absence of symptoms, 1 = Mild symptoms, 2 = Moderate symptoms and 3 = Severe symptoms. The scores of each individual symptom (runny nose, blocked nose and the maximum score of nasal itching or sneezing) will be added together to give a TNSS of 0 to 9. TNSS Score 0 indicates better outcome and TNSS score 9 indicates worse outcome.
  Number of Participants Analyzed is based on all patients with evaluable efficacy and/or biomarker data at visit 11.
Time Frame: Pre-dose on visit 11 (end of 3rd week of treatment)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | AZD8848 20 μg x3 | Placebo | AZD8848 60 μg
Number analyzed (Participants) | 49 | 15 | 15
Scores on a scale | 1.20 (1.020) | 0.67 (1.047) | 0.80 (0.862)

11. Secondary Outcome: Absolute Mean Value of Peak Nasal Inspiratory Flow (PNIF)
Description: Absolute mean value of Peak Nasal Inspiratory Flow (PNIF) for pre-dose symptoms on visit 2, during treatment period. Treatment period is one month, which starts at visit 2 and ends at visit 14. The patient will breathe out as much as he can. Then a mask (Portable Inspiratory Flow Meter) will be placed over the nose and mouth and the patient will inspire forcefully through the nose while the lips remain tightly closed. The highest PNIF (L/minute) out of 3 measurements will be recorded.
  Number of Participants Analyzed is based on all patients with evaluable efficacy and/or biomarker data at visit 2.
Time Frame: Pre-dose on visit 2 (baseline)
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | AZD8848 20 μg x3 | Placebo | AZD8848 60 μg
Number analyzed (Participants) | 50 | 16 | 17
L/min | 170.4 (54.593) | 176.9 (63.005) | 169.4 (62.497)

12. Secondary Outcome: Absolute Mean Value of Peak Nasal Inspiratory Flow (PNIF)
Description: Absolute mean value of Peak Nasal Inspiratory Flow (PNIF) for pre-dose symptoms on visit 11, during treatment period. Treatment period is one month, which starts at visit 2 and ends at visit 14. The patient will breathe out as much as he can. Then a mask (Portable Inspiratory Flow Meter) will be placed over the nose and mouth and the patient will inspire forcefully through the nose while the lips remain tightly closed. The highest PNIF (L/minute) out of 3 measurements will be recorded.
  Number of Participants Analyzed is based on all patients with evaluable efficacy and/or biomarker data at visit 11.
Time Frame: Pre-dose on visit 11 (end of 3rd week of treatment)
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | AZD8848 20 μg x3 | Placebo | AZD8848 60 μg
Number analyzed (Participants) | 49 | 15 | 15
L/min | 168.1 (52.070) | 191.3 (48.824) | 182.7 (61.350)

13. Secondary Outcome: Change From Baseline of C-X-C Motif Chemokine 10 (CXCL10) in Plasma
Description: Change from baseline to 24 hours after last dose (day1 visit 15) of C-X-C motif chemokine 10 (CXCL10) in plasma, expressed as a ratio. The ratio is calculated as day1 of visit 15 / baseline.
  Number of Participants Analyzed is based on all patients with evaluable biomarker data at visit 2 and visit15.
Time Frame: Baseline to 1st day of visit 15
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD8848 20 μg x3 | Placebo | AZD8848 60 μg
Number analyzed (Participants) | 46 | 15 | 16
ratio | 2.89 [2.45 to 3.40] | 0.803 [0.6 to 1.07] | 3.90 [2.96 to 5.15]

14. Secondary Outcome: Change From Baseline of C-X-C Motif Chemokine 10 (CXCL10) in Nasal Lavage
Description: Change from baseline to 24 hours after last dose (day1 visit 15) of C-X-C motif chemokine 10 (CXCL10) in nasal lavage, expressed as a ratio. The ratio is calculated as day1 of visit 15 / baseline.
  Number of Participants Analyzed is based on all patients with evaluable biomarker data at visit 2 and visit 15.
Time Frame: Baseline to 1st day of visit 15
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | AZD8848 20 μg x3 | Placebo | AZD8848 60 μg
Number analyzed (Participants) | 48 | 14 | 15
ratio | 30.0 [21.99 to 40.81] | 1.66 [0.93 to 2.97] | 26.9 [15.52 to 46.56]

ADVERSE EVENTS:
Arm/Group | AZD8848 20 μg x3 | Placebo | AZD8848 60 μg
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 48/50 | 12/16 | 12/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD8848 20 μg x3 (N=50) | Placebo (N=16) | AZD8848 60 μg (N=17)
Eye Pruritus (Eye disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1 | 1
Asthenia (General disorders) | 4 | 0 | 1
Chills (General disorders) | 6 | 0 | 3
Fatigue (General disorders) | 7 | 1 | 1
Feeling abnormal (General disorders) | 3 | 0 | 1
Irritability (General disorders) | 0 | 0 | 1
Pain (General disorders) | 3 | 1 | 3
Pyrexia (General disorders) | 11 | 0 | 1
Nasopharyngitis (Infections and infestations) | 5 | 2 | 0
Sinusitus (Infections and infestations) | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0
Disgeusia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 20 | 5 | 3
Migraine (Nervous system disorders) | 0 | 0 | 1
Stress (Psychiatric disorders) | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 24 | 1 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 | 1 | 4
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 17 | 3 | 6
Sneezing (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 14 | 3 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 4 | 9
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Scab (Skin and subcutaneous tissue disorders) | 4 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 0 | 1
Herpes Virus Infection (Infections and infestations) | 3 | 0 | 0
Eczema Eyelids (Eye disorders) | 0 | 1 | 0
Eye Oedema (Eye disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between PI and Sponsor (AZ) or its agents that restricts the PI's right to discuss/publish trial results after the trial is completed. The PI agrees to collaborate in good faith with AZ with regards to content and formation of any publication or disclosure to be made by PI and to pay due consideration to opinions offered by AZ